CLINICAL TRIAL: NCT05943418
Title: Examining the Effectiveness of Wysa's Computerized Cognitive Behavioral Therapy Program (a Digital Mental Health Intervention) in Reducing Symptoms of Anxiety: Randomized Control Trial
Brief Title: Examining the Effectiveness of Wysa for Worry Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wysa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Wysa_RCT_01
Record Dates: First submitted 2023-06-19; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Anxiety
Keywords: Worry; Anxiety; Digital Mental Health
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial with an intervention arm and a control arm.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention (Experimental)
  Interventions: Behavioral: Wysa for Worry
- Control arm (Active Comparator)
  Interventions: Behavioral: App-based Psychoeducation

INTERVENTIONS:
Behavioral: Wysa for Worry — The Wysa for Worry cCBT program is a week-based cCBT programme consisting of specialised cognitive behavior therapy (CBT) interventions delivered through a conversational agent.
  Each week of the programme focuses on a different CBT technique or intervention, which is explained in a short weekly video. Following each video, the technique or intervention is discussed and practiced with Wysa's AI chatbot.
  Arms: Active Intervention
Behavioral: App-based Psychoeducation — The control will include the weekly delivery of active psychoeducational resources.
  Arms: Control arm

SUMMARY:
The goal of this randomized controlled trial is to test for the effectiveness of Wysa's Worry computerized cognitive behaviour therapy (cCBT) program (a digital mental health intervention) in comparison to a digital app that offers psychoeducation to patients who have mild to moderate symptoms of anxiety.

DETAILED DESCRIPTION:
People dealing with worry can receive augmented support from digital mental health interventions. The intervention being tested in this study is Wysa's Worry cCBT program. Its outcomes will be compared to a randomized, controlled arm that offers psychoeducation.

For the purpose of this study participants will be recruited through different online channels and will be randomly assigned to either the intervention or control group. Regardless of their assignment they will be completing weekly standardized assessments examining their symptoms of anxiety and depression, and examining any improvement.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the study is as follows:

  * Patients who are at least 18 years of age.
  * Patients who have mild to moderate symptoms of anxiety (scores: 5-15, according to GAD-7).
  * Patients who are not already engaged in psychological therapy and not intending to start psychological therapy in the next eight weeks.
  * Patients who haven't used any DMHI (Digital Mental Health Interventions) in the last 6 months.
  * Patients without risk of suicidal ideation and behaviour.
  * Patients who are capable of reading and understanding English and have provided written or verbal informed consent to participate.
  * Patients who own and use a smartphone with functional audio.

Exclusion Criteria:

* Patients who are at an increased risk of suicide.
* Patients with diagnosis of or receiving treatment for alcohol/substance use disorder.
* Patients who've had their psychiatric medication or dose changed in the last 1 month.
* Patients who suffer from severe anxiety
* Patients with diagnosis of or receiving treatment for an active state of psychosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in scores of Generalized Anxiety Disorder Scale (GAD-7) | Baseline, Weekly assessments for 7 weeks, Post intervention assessment (one month after the participant finishes the intervention)
  GAD-7 is a 7 item assessment that screens for anxiety and assesses the severity of anxiety symptoms.

SECONDARY OUTCOMES:
Change in scores of Patient Health Questionnaire-9 (PHQ-9) | Baseline, Weekly assessments for 7 weeks, Post intervention assessment (one month after the participant finishes the intervention)
  PHQ-9 is a 9 item assessment that screens for depressive symptoms and assesses the severity of the depressive symptoms.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with any external party as it does not comply with the terms of consent.

REFERENCES:
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941